CLINICAL TRIAL: NCT02443701
Title: Low Level Laser Therapy and Neuromuscular Electrical Stimulation on Knee Extension Strength and Jump in Volleyball Athletes: a Randomized Controlled Trial
Brief Title: Light Therapy and Electrical Stimulation on Functional Performance in Volleyball Athletes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centro de Traumatologia do Esporte (Other)
Responsible Party: Principal Investigator, Ronaldo A Cunha, PT, Coordinator, Centro de Traumatologia do Esporte
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: U1111-1169-4661
Record Dates: First submitted 2015-04-23; First posted 2015-05-14 (Estimated); Last update posted 2015-08-13 (Estimated); Status verified 2015-08

CONDITIONS: Muscle Weakness; Sports Performance
MeSH Terms: conditions — Muscle Weakness | interventions — Exercise; Plyometric Exercise; Lasers; Phototherapy

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Exercise (Experimental): All 12 volleyball athletes performed a strength training and jump, to be held in both legs at the same time. The training will be held in a six-week period, a total of 18 training. Athletes will hold a warmup in stationary bike for 6 minutes, maximum isometric strengthening in leg extension (knee positioned at 60 ° of flexion and hip in 75 ° of flexion), 10 repetitions of 10 seconds with 30 seconds interval. After strengthening conduct a complete rest 5 minutes and jump training countermovement in 5 sets of 10 jumps (1 minute interval between each jump).
  Interventions: Other: Exercise
- NEMES (Experimental): All 12 volleyball athletes performed a strength training and jump, to be held in both legs at the same time. The training will be held in a six-week period, a total of 18 training. Athletes will hold a warmup in stationary bike for 6 minutes, maximum isometric strengthening in leg extension (knee positioned at 60 ° of flexion and hip in 75 ° of flexion), 10 repetitions of 10 seconds with 30 seconds interval. After strengthening conduct a complete rest 5 minutes and jump training countermovement in 5 sets of 10 jumps (1 minute interval between each jump).The healthy athletes electrical stimulation group will perform the same training program described above, but strength training is associated with electrical stimulation, medium frequency current (1kHz), modulated at 70Hz, cycle Work 10%, intensity used will vary according to the capacity and tolerable for each individua. The stimulated muscle group will be the quadriceps femoris
  Interventions: Other: Exercise; Other: NMES
- Phototherapy (Experimental): All 12 volleyball athletes performed a strength training and jump, to be held in both legs at the same time. The training will be held in a six-week period, a total of 18 training. Athletes will hold a warmup in stationary bike for 6 minutes, maximum isometric strengthening in leg extension (knee positioned at 60 ° of flexion and hip in 75 ° of flexion), 10 repetitions of 10 seconds with 30 seconds interval. After strengthening conduct a complete rest 5 minutes and jump training countermovement in 5 sets of 10 jumps (1 minute interval between each jump). The 12 healthy athletes participating in the phototherapy group will undergo a phototherapy protocol before performing the strength and jump training. Phototherapy will be conducted through a cluster with 03 diodes with 850nm wavelength and the following parameters: Power 50mW diode, diode energy by 2J. The application sites will be six points on the belly of the quadriceps femoris muscles bilaterally.
  Interventions: Other: Exercise; Other: LASER

INTERVENTIONS:
Other: Exercise — Warmup program, maximum isometric strengthening, and jump training
  Other Names: Plyometric training
Other: LASER — a cluster with 03 diodes with 850nm wavelength and the following parameters: Power 50mW diode, diode energy by 2J, power per point of 6J, totaling 36J per member
  Other Names: Phototherapy
  Arms: Phototherapy
Other: NMES — electrical stimulation, medium frequency current (1kHz), Burst duration equal to 2ms with, modulated at 70Hz, cycle Work 10% T-on and T-10 seconds off and 30 seconds intensity used will vary according to the capacity and tolerable for each individual
  Arms: NEMES

SUMMARY:
Background: Volleyball players constantly perform vertical jumps, the higher the height of the jump is better sports performance of these players. Several methods have been tested to improve jumping performance in these players. It will be investigated the addition of electrical stimulation and phototherapy to jump training in volleyball athletes. DESIGN: randomized controlled trial. METHODS: This study will be conducted with 36 male athletes volleyball with minimum experience of 12 months sport. Will be randomized and assigned to 3 groups (control group, NEMES group and group phototherapy). All 36 healthy volleyball athletes who passed the initial selection and agreed to participate in the study, conduct a muscle strength and jump training program, which is held in both legs simultaneously. The 12 healthy athletes electrical stimulation group will perform the same training program described above, but strength training is associated with electrical stimulation. The 12 healthy athletes participating in the phototherapy group will undergo a phototherapy protocol before performing the strength and jump training. All selected participants will undergo an assessment of muscle strength of knee extensors and evaluate the jump. These evaluations were baseline, 6 weeks and 8 weeks after baseline.

DETAILED DESCRIPTION:
Background: Volleyball players constantly perform vertical jumps, the higher the height of the jump is better sports performance of these players. Several methods have been tested to improve jumping performance in these players. It will be investigated the addition of electrical stimulation and phototherapy to jump training in volleyball athletes.

DESIGN: randomized controlled trial METHODS This study will be conducted with 36 male athletes volleyball with minimum experience of 12 months sport. Will be randomized and assigned to 3 groups (control group, NEMES group and group phototherapy).INTERVENTION All 36 healthy volleyball athletes who passed the initial selection and agreed to participate in the study, conduct a muscle strength and jump training program, which is held in both legs simultaneously. The training will be held in a period of six weeks with frequency of three times a week, totaling 18 training. The interval between one session and another will be 24 hours.

STRENGTH TRAINING To conduct the training all 36 healthy athletes, carry out heating in stationary bike for six minutes. After heating, the individuals are positioned in the extension machine with the knee joint positioned at 60 ° of flexion and hip at 75 ° flexion, which will perform 10 repetitions of maximal voluntary isometric contraction (MVIC), and the isometric contraction time will be 10 seconds and the rest time between repetitions of 30 seconds.

JUMPING TRAINING After the training the leg extension 36 individuals remain at rest for 5 minutes before starting the jump training. One type of jumps will be trained, countermovement jump (SCM). SCM in the participant will begin the movement of an upright standing position, with the knees fully extended, the volunteer will bend your knees up to about 90 ° before starting the movement up the jump. In each jump training individuals hold five sets of 10 repetitions with one minute intervals between each series.

ELECTRICAL STIMULATION The 12 healthy athletes electrical stimulation group will perform the same training program described above, but strength training is associated with electrical stimulation, medium frequency current (1kHz), Burst duration equal to 2ms with, modulated at 70Hz, cycle Work 10% T-on and T-10 seconds off and 30 seconds intensity used will vary according to the capacity and tolerable for each individual will be recorded for later analysis. The stimulated muscle group will be the quadriceps muscle, with two self-adhesive electrodes 8x13 cm (area of 104cm2). An electrode is placed in the rectus femoris muscle region with a distance of 20 cm from the anterior superior iliac crest and the other is positioned on the oblique vastus muscle region with a distance of 5 cm from the superior pole of the patella.

PHOTOTHERAPY The 12 healthy athletes participating in the phototherapy group will undergo a phototherapy protocol before performing the strength and jump training. Phototherapy will be conducted through a cluster with 03 diodes with 850nm wavelength and the following parameters: Power 50mW diode, diode energy by 2J, power per point of 6J, totaling 36J per member. The irradiation time is 40s by point in the continuous mode. The laser is applied in stationary manner in touch and perpendicular to the skin. The application sites will be six points on the belly of the quadriceps muscles bilaterally.

Evaluation and monitoring All selected participants will undergo an assessment of muscle strength of knee extensors and evaluate the jump. These evaluations were baseline, 6 weeks and 8 weeks after baseline.

The maximum isometric muscle strength of the knee extensors will be quantified using a hand dynamometer. To evaluate the ability of the jump was performed Jump and Reach Test. The maximum amount of countermovement jumps will be performed for 2 minutes. The overall impression will be assessed by scale of perceptation of the overall effect.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers;
* volleyball players;
* gender male;
* non-smoking;
* aged between 17 and 18;
* weight within 15% variation limit of normal weight for male athletes, taking into account height and physique.

Exclusion Criteria:

* smoking volunteers;
* history of alcohol or substance abuse;
* diagnosis of cardiac, renal, gastrointestinal, hepatic, pulmonary, neurological, psychiatric, hematological or metabolic disorders; that are not available to participate in all stages of the study.

Ages: 17 Years to 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 36 (Estimated)
Dates: Start 2015-07; Primary Completion 2015-07 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Muscle strength measured by dynamometer | 6 weeks
  The athletes will be evaluated in 3 phases: initial evaluation (pre-training), immediately after post-training, and a 8-wk follow up. It will be assessed the isometric muscle strength of knee extensors.

SECONDARY OUTCOMES:
Global impression measured by global perceived effect scale | 6 weeks
  The athletes will be evaluated in 3 phases: initial evaluation (pre-training), immediately after post-training, and a 8-wk follow up. It will be assessed the global perceived effect scale about the jump.
Jumping frequency measured by jumping frequency in 2 minutes | 6 weeks
  The athletes will be evaluated in 3 phases: initial evaluation (pre-training), immediately after post-training, and a 8-wk follow up. It will be assessed Jumping frequency in 2 Minutes (countermovement jump)
Jump ability measured by jump ability test | 6 weeks
  The athletes will be evaluated in 3 phases: initial evaluation (pre-training), immediately after post-training, and a 8-wk follow up. It will be assessed the jump ability test.

CONTACTS AND LOCATIONS:
Locations (1):
- Ronaldo Alves da Cunha, São Paulo, São Paulo, Brazil